CLINICAL TRIAL: NCT00355654
Title: Safety and Immunogenicity of Booster Vaccination With PEDIACEL®, a Combined Diphtheria, Tetanus, Five Component Acellular Pertussis, Inactivated Poliomyelitis and Haemophilus Influenzae Type b Conjugate Vaccine (Adsorbed), Compared to Booster Vaccination With Infanrix® Hexa When Both Vaccines Are Co-Administered With Prevenar® to Toddlers 11-18 Months of Age
Brief Title: Study to Compare Booster Vaccination With Pediacel® to Infanrix® Hexa When Both Are Co-Administered With Prevenar®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A5I19
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Infant; Healthy
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Haemophilus influenzae type b; Hepatitis B
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections; Hepatitis B | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Participants will receive PEDIACEL with Prevenar at Visit 1 and ENGERIX-B Kinder at Visit 2
  Interventions: Biological: DT5aP-IPV-Hib 5-component Pertussis vaccine
- Group 2 (Active Comparator): Participants will receive Infanrix hexa with Prevenar at Visit 1
  Interventions: Biological: DT3aP-HBs-IPV

INTERVENTIONS:
Biological: DT5aP-IPV-Hib 5-component Pertussis vaccine — 0.5 mL, IM
  Other Names: Pediacel™
  Arms: Group 1
Biological: DT3aP-HBs-IPV — 0.5 mL, IM
  Other Names: Infanrix® hexa
  Arms: Group 2

SUMMARY:
The purpose of the study is to provide data on the safety and immunogenicity of Pediacel® to allow its use as a fourth dose administered to 11-18 months old toddlers at the same time as Prevenar®.

Primary Objective:

To evaluate the safety of Pediacel® booster dose co-administered with Prevenar® to toddlers at 11-18 months of age.

Secondary Objectives:

* To describe the incidence rate of severe fever within four days post-vaccination
* To describe the antibody responses to all antigens in a subgroup of subjects at baseline and post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers 11-18 months of age (from the 11th month birthday to one day prior to the 19th month birthday) who previously received the primary immunisation series with a hexavalent vaccine (consisting of three doses of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B and Haemophilus influenza type b combined vaccine administered within the first 6 months of life)
* Informed consent form signed by both parents or by the legal guardian
* Parents or a legal guardian able to read and write the local language
* Parents or a legal guardian able to attend all scheduled visits and to comply with the study procedures.

Exclusion Criteria:

* Presence of fever (defined as rectal body temperature ≥ 38.0°C) reported within the last 72 hours
* Moderate or severe acute illness with or without fever
* Participation in another clinical trial in the 30 days preceding study vaccination
* Planned participation in another clinical trial during the present study period
* Immunisation with a pneumococcal vaccine prior to study vaccination or planned during the participation in the study
* Received more than 3 doses of a hexavalent vaccine prior to study vaccination
* Received any vaccination in the 30 days preceding the trial
* History of serological/microbiologically-confirmed diagnosis of infection due to pertussis, tetanus, diphtheria, poliomyelitis, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae
* Congenital or acquired humoral/cellular immunodeficiency or immunosuppressive therapy such as long-term systemic corticosteroids therapy (≥ 2 mg/kg/day prednisone equivalent for ≥ 14 days in the 30 days prior to study vaccination)
* Systemic or local hypersensitivity to any of the study vaccine components (including neomycin, streptomycin, polymyxin B and formaldehyde)
* History of a life-threatening reaction (such as encephalopathy, Hypotonic-Hyporesponsive Episode (HHE), rectal body temperature ≥ 40.0°C, convulsions with or without fever) to any vaccine containing the same components as the study vaccines
* Blood or blood-derived products (immunoglobulins) received during 3 months prior to study vaccination
* Known HIV seropositivity
* Known thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of encephalopathy, seizures or progressive, evolving or unstable neurological condition
* Clinically significant findings on review of systems that might interfere with study vaccination or which, in the opinion of the Investigator, would interfere with the evaluation of the study vaccine/objectives or pose a health risk to the subject.

Ages: 11 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 847 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety after administration of PEDIACEL® booster dose | 0 to 3 Days post-vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety (as fever rate) after administration of PEDIACEL® Vaccine | 4 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (69):
- Germany (69):
  - Aalen
  - Aisch
  - Alsfeld
  - Augsburg
  - Bad Oeynhausen
  - Bad Säckingen
  - Berlin
  - Bernau B. Berlin
  - Bielefeld
  - Bönnigheim
  - Bramsche
  - Bretten
  - Cham
  - Cologne
  - Datteln
  - Detmold
  - Eisenberg
  - Erfurt
  - Espelkamp
  - Frankenthal
  - Freiburg im Breisgau
  - Gerolstein
  - Gersthofen
  - Goch
  - Göttingen
  - Gütersloh
  - Hamburg
  - Hechtsheim
  - Herbolzheim
  - Herrsching am Ammersee
  - Jena
  - Karlsruhe
  - Karlstadtm
  - Kehl
  - Kempten
  - Korbach
  - Königstein/Taunus
  - Krefeld
  - Landshut
  - Lauf/Pegnitz
  - Lauffen am Neckar
  - Leinfelden-Echte
  - Lindenberg
  - Lingen 49 (Ems)
  - Ludwigshafen
  - Magdeburg
  - Mainz
  - Mannheim
  - Marburg
  - Marktoberdorf
  - Marktredwitz
  - Melle
  - Mönchengladbach
  - München
  - Nabburg
  - Neumünster
  - Niedernhausen
  - Prüm
  - Schwäbisch Gmünd
  - Schwäbisch Hall
  - Schwieberdingen
  - Solingen
  - Traunreut
  - Ulm
  - Unterschleissheim
  - Weinheim
  - Wiesbaden
  - Wildeshausen
  - Wolfenbüttel

REFERENCES:
- [Derived] Berner R, Boisnard F, Thomas S, Mwawasi G, Reynolds D. Safety and immunogenicity of fully liquid DTaP(5)-IPV-Hib pediatric combination vaccine (Pediacel(R)) compared to DTaP(3)-HBV-IPV/Hib (Infanrix(R) Hexa) when coadministered with heptavalent pneumococcal conjugate vaccine (PCV7) as a booster at 11-18 months of age: a phase III, modified double-blind, randomized, controlled, multicenter study. Vaccine. 2012 Jul 27;30(35):5270-7. doi: 10.1016/j.vaccine.2012.05.064. Epub 2012 Jun 9. PMID 22691430
- See also: Related Info — http://www.sanofipasteur.com